CLINICAL TRIAL: NCT06060041
Title: IC-8 Apthera IOL New Enrollment Post Approval Study
Status: Recruiting | Type: Observational
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: SAIL-101-PAS2
Record Dates: First submitted 2023-09-19; First posted 2023-09-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cataract; Presbyopia; Posterior Capsule Opacification
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IC-8 Apthera intraocular lens (IOL) Group: Patients previously implanted with the IC-8 Apthera intraocular lens (IOL) and who have developed posterior capsular opacification (PCO) which requires treatment with Nd:YAG laser capsulotomy.

SUMMARY:
The purpose of this study is to verify the post-market safety of the IC-8 Apthera IOL after the treatment of posterior capsular opacification (PCO), an expected complication related to IC-8 Apthera IOL implantation.

DETAILED DESCRIPTION:
Prospective, multi-center, single-group, non-randomized new enrollment post approval study to assess the post-market safety of the IC-8 Apthera IOL after Nd:YAG laser capsulotomy following sufficient surgeon training of the sponsor-recommended standardized Nd:YAG laser capsulotomy technique. All subjects will undergo approximately 6 study visits and will be followed 24 months post IC-8 Apthera IOL implantation. There is one study group: subjects previously implanted with the IC-8 Apthera IOL and who have developed posterior capsular opacification (PCO) which requires treatment with Nd:YAG laser capsulotomy.

ELIGIBILITY:
Inclusion Criteria:

* 22 years of age or older, any race and any gender;
* Posterior capsule opacification (PCO) requiring treatment in the IC-8 Apthera IOL eye
* Able to comprehend and have signed a statement of informed consent;
* Availability, willingness, ability and sufficient cognitive awareness to comply with examination procedures and study visits;
* Clear intraocular media in both eyes;
* Preoperative corneal astigmatism ≤1.5 D in the IC-8 Apthera IOL eye prior to IC-8 Apthera implantation;
* Prior IC-8 Apthera IOL implantation in one eye and a monofocal/monofocal toric IOL in the other eye in accordance with the directions for use (DFU) for each IOL.

Exclusion Criteria:

* Pharmacologically dilated pupil size less than 7.0 mm in the IC-8 Apthera IOL eye;
* Irregular astigmatism in either eye;
* History of retinal disease;
* Active or recurrent anterior segment pathology;
* Presence of ocular abnormalities;
* Diagnosis of dry eye in which patients are unable to maintain eye comfort or adequate vision even with dry eye treatment;
* Previous corneal or intraocular surgery, except cataract surgery;
* History of ocular trauma or ocular conditions expected to require retinal laser treatment or other surgical intervention;
* Acute, chronic or uncontrolled systemic disease that would, in the opinion of the investigator, confound the outcomes of the study;
* Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with hormonal fluctuation that could lead to refractive changes and dry eye;
* Concurrent participation or participation in any clinical trial up to 30 days prior to the first visit in the study.
* Subjects who plan to be traveling, relocating or otherwise unavailable to attend any of the visits

Min Age: 22 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Potential study subjects will be recruited from patients previously implanted with the IC-8 Apthera intraocular lens (IOL) and who have developed posterior capsular opacification in the IC-8 Apthera IOL eye which requires treatment with Nd:YAG laser capsulotomy
Sampling Method: Non-Probability Sample
Enrollment: 435 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of any additional Nd:YAG laser treatments beyond the initial Nd:YAG laser treatment | 24 Months post IC-8 Apthera IOL Implantation
  Rates of additional Nd:YAG laser treatments in the eye implanted with the IC-8 Apthera intraocular lens (IOL) beyond the initial Nd:YAG laser treatment will be assessed through 24 months post IC-8 Apthera IOL implantation
Nd:YAG laser treatment outcome and/or complications | 24 Months post IC-8 Apthera IOL Implantation
  Nd:YAG laser treatment outcomes and/or complications in the eye implanted with the IC-8 Apthera intraocular lens (IOL) will be assessed through 24 months post IC-8 Apthera IOL implantation.
IOL related assessments | 24 Months post IC-8 Apthera IOL implantation
  The appearance of the IC-8 Apthera intraocular lens (IOL) will be assessed through 24 months post IC-8 Apthera IOL implantation
Rates of Secondary Surgical Interventions (SSIs) | 24 Months post IC-8 Apthera IOL implantation
  Rates of secondary surgical interventions in the IC-8 Apthera intraocular lens (IOL) eyes and the fellow eyes will be assessed through 24 months post IC-8 Apthera IOL implantation
Rates of other serious adverse events | 24 Months post IC-8 Apthera IOL implantation
  Rates of other serious adverse events in the IC-8 Apthera intraocular lens (IOL) eyes and fellow eyes will be evaluated through 24 months post IC-8 Apthera IOL implantation
Rates of ocular adverse events | 24 Months post IC-8 Apthera IOL implantation
  Rates of ocular adverse events in the IC-8 Apthera intraocular lens (IOL) eyes and fellow eyes will be evaluated through 24 months post IC-8 Apthera IOL implantation
Rates of subjective visual disturbances per the Quality of Vision (QoV) Questionnaire | 24 Months post IC-8 Apthera IOL implantation
  Subjective responses to the QoV Questionnaire that assess frequency of visual disturbances (from 'never' to 'very often'), severity of those disturbances (from 'not at all' to 'severe') and bothersomeness of those disturbances (from 'not at all' to 'very') in both the IC-8 Apthera intraocular lens (IOL) eyes and the fellow eyes.
Rates of subjective visual disturbances per the Small Aperture Patient Questionnaire (SAPQ) | 24 Months post IC-8 Apthera IOL implantation
  Subjective responses to the Small Aperture Patient Questionnaire (SAPQ) that assess frequency of visual disturbances (from 'never' to 'very often'), severity of those disturbances (from 'not at all' to 'severe') and bothersomeness of those disturbances (from 'not at all' to 'very') in both the IC-8 Apthera intraocular lens (IOL) eyes and the fellow eyes.

OTHER OUTCOMES:
Nd:YAG laser technique details and/or settings | PCO treatment visit (during the Nd:YAG laser procedure)
  Nd:YAG laser technique and/or settings during treatment in an IC-8 Apthera intraocular lens (IOL) eye will be evaluated
Investigator opinion of ease of YAG procedure | PCO treatment visit (during the Nd:YAG laser procedure)
  Difficulty performing Nd:YAG laser treatment in an IC-8 Apthera intraocular lens (IOL) eye will be evaluated per scale of difficulty chosen by investigator from 'No difficulty' to 'Great difficulty'
Mean monocular and binocular uncorrected distance visual acuity (UCDVA), uncorrected intermediate visual acuity (UCIVA) and uncorrected near visual acuity (UCNVA) | 24 Months post IC-8 Apthera IOL implantation
  Mean monocular and binocular uncorrected distance visual acuity (UCDVA), uncorrected intermediate visual acuity (UCIVA) and uncorrected near visual acuity (UCNVA) will be evaluated in the IC-8 Apthera intraocular lens (IOL) eyes and the fellow eyes (same units of measure for all measurements)
Mean monocular and binocular distance corrected distance visual acuity (DCDVA), distance corrected intermediate visual acuity (DCIVA) and distance corrected near visual acuity (DCNVA) | 24 Months post IC-8 Apthera IOL implantation
  Mean monocular and binocular distance corrected distance visual acuity (DCDVA), distance corrected intermediate visual acuity (DCIVA) and distance corrected near visual acuity (DCNVA) will be evaluated in the IC-8 Apthera intraocular lens (IOL) eyes and the fellow eyes (same units of measure for all measurements)
Rates of device deficiencies | 24 Months post IC-8 Apthera IOL implantation
  Rates of device deficiencies in the IC-8 Apthera intraocular lens (IOL) eyes and the fellow eyes will be evaluated
Rates of loss of 10 or more Early Treatment Diabetic Retinopathy Study (ETDRS) letters of best corrected distance visual acuity (BCDVA) | 24 Months post IC-8 Apthera IOL implantation
  The rates of each event of loss of 10 or more Early Treatment Diabetic Retinopathy Study (ETDRS) letters of best corrected distance visual acuity (BCDVA) between a study visit and a later study visit, the reason for the visual acuity loss, and the treatment/outcome of these instances will be assessed through 24 months post IC-8 Apthera intraocular lens (IOL) implantation

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Trinity Research Group, LLC, Dothan, Alabama
  - Feinerman Vision Center, Newport Beach, California
  - Argus Research Center, Cape Coral, Florida
  - Stephenson Eye Associates, Venice, Florida
  - Virdi Eye Clinic and Laser Vision Center, Rock Island, Illinois
  - Price Vision Group, Indianapolis, Indiana
  - Grene Vision Group, Wichita, Kansas
  - Oakland Eye, Birmingham, Michigan
  - Vance Thompson Vision - Omaha, Omaha, Nebraska
  - Eye Associates of New Jersey, Dover, New Jersey
  - Northern New Jersey Eye Institute, South Orange, New Jersey
  - Ophthalmic Partners, PC, Bala-Cynwyd, Pennsylvania
  - Berkeley Eye Center, Sugar Land, Texas
  - Utah Eye Centers, Bountiful, Utah

IPD SHARING:
Plan to Share IPD: No